CLINICAL TRIAL: NCT01114529
Title: A 24-month, Multi-center, Open-label, Randomized, Controlled Trial to Investigate Efficacy, Safety and Evolution of Cardiovascular Parameters in de Novo Renal Transplant Recipients After Early Calcineurin Inhibitor to Everolimus Conversion
Brief Title: Efficacy, Safety and Evolution of Cardiovascular Parameters in Renal Transplant Recipients
Acronym: ELEVATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2429; 2009-015918-22 (EudraCT Number)
Record Dates: First submitted 2010-04-27; First posted 2010-05-03 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Kidney Transplantation
Keywords: de novo renal allograft recipients; renal allograft function; CNI-free regimen
MeSH Terms: interventions — Everolimus; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Experimental): Conversion from CNI to everolimus in combination with Myfortic and steroids
  Interventions: Drug: Everolimus
- Calcineurin inhibitor, Prograf or Neoral (Active Comparator): Control arm: CNI continuation, either Prograf or Neoral in combination with Myfortic and steroids
  Interventions: Drug: Prograf or Neoral

INTERVENTIONS:
Drug: Everolimus — Early CNI to everolimus conversion
  Other Names: Certican, Zortress, RAD001
  Arms: Everolimus
Drug: Prograf or Neoral — Active CNI-based control (Prograf or Neoral)
  Other Names: Tacrolimus or Cyclosporine
  Arms: Calcineurin inhibitor, Prograf or Neoral

SUMMARY:
The purpose of this study was to determine whether an early Calcineurin Inhibitor (CNI) to everolimus conversion at 10-14 weeks post transplantation improves renal allograft function without compromising efficacy compared to standard CNI treatment in de novo renal allograft recipients. In addition, the study was designed to evaluate the impact of a CNI-free regimen on evolution of cardiovascular parameters in de novo renal allograft recipients

DETAILED DESCRIPTION:
This was a 24-month, multi-center, randomized, open-label trial with two parallel arms in adult de novo renal allograft recipients. The study consisted of a run-in period from transplantation to Randomization and a treatment period from Randomization until Month 24. At baseline visit, patients were transplanted and entered the run-in period from transplantation (Baseline) to Randomization (week 10-14 post-transplantation). At Week 10-14, eligible patients were randomized into one of the 2 treatment arms: standard CNIs and Myfortic versus everolimus and Myfortic and entered the treatment period of the study from Randomization to Month 24. Patients in both arms received steroids as per center practice and in any caseat least 5 mg/Day. At Randomization, patients were stratified according to their renal allograft function and previous cardiovascular events. The main analysis was performed at Month 12 and the follow-up analysis was performed at Month 24.

ELIGIBILITY:
Inclusion Criteria at Baseline:

* Male or female renal allograft recipients at least 18 years old.
* Written informed consent.
* Patient receiving a primary or secondary kidney transplant from a cadaveric or living unrelated-/related donor.
* Cold ischemia time (CIT) < 24 hours.
* Negative pregnancy test for female patients.

Inclusion Criteria at Randomization:

* Patients on CNI (TAC or CsA) + Myfortic + steroids.
* Serum creatinine < 2.8 mg/dL (250 µmol/L) and an actual eGFR (MDRD4) ≥ 25 mL/min/1.73m exp2 (without renal replacement therapy).

Exclusion Criteria at Baseline:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

* Recipient of multiple organ transplants.
* Recipient of ABO incompatible allograft or a positive cross-match.
* Panel Reactive Antibodies (PRA) level ≥ 30 %.
* Positive test for human immunodeficiency virus (HIV).
* Patient receiving an allograft from a Hepatitis B surface Antigen (HBsAg) or a Hepatitis C Virus (HCV) positive donor.
* HBsAg and/or a HCV positive patient with evidence of elevated LFTs (ALT/AST levels ≥ 2.5 times ULN).
* Severe restrictive or obstructive pulmonary disorders.
* Patient with severe allergy requiring acute or chronic treatment or hypersensitivity to any of the study drugs or similar drugs.
* Severe hypercholesterolemia or hypertriglyceridemia.
* Low platelet count.
* Low white blood cell count.
* History of malignancy of any organ system

Exclusion Criteria at Randomization:

* Graft loss.
* Patient on renal replacement therapy.
* Patient who experienced severe humoral and/or cellular rejection (BANFF ≥ IIb).
* Patient with ≥ 2 episodes of AR or an AR episode that needed antibody treatment.
* Patient with ongoing or currently treated AR (2 weeks prior to randomization).
* Proteinuria > 1 g/day.
* Patients with recurrence of Focal Segmental Glomerulosclerosis (FSGS).
* Low platelet count; Low white blood cell count; Low absolute neutrophil count; Low hemoglobin.
* Severe liver disease.
* Systemic infection requiring continued therapy that would interfere with the objectives of the study.
* Severe hypercholesterolemia or hypertriglyceridemia.
* Patients with ongoing wound healing problems, clinically significant infection requiring continued therapy.
* Presence of intractable immunosuppressant complications or side effects.
* Patients on anticoagulants that prevents renal allograft biopsy.
* Use of prohibited medication.
* Use of immunosuppressive agents not utilized in the protocol.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential not using a highly effective method of birth control.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2010-08-09 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2014-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (71):
- Argentina (5):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, Resistencia, Chaco Province
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Santa Fe
- Australia (4):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Tartu, Estonia
- France (5):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (8):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hannover Muenden
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Münster
- Greece (2):
  - Novartis Investigative Site, Pátrai, Greece
  - Novartis Investigative Site, Athens
- India (5):
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, New Delhi
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Riga, Latvia
- Novartis Investigative Site, Vilnius, Lithuania
- Mexico (4):
  - Novartis Investigative Site, Torreón, Coahuila
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Veracruz
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leiden
- Novartis Investigative Site, Oslo, Norway
- Portugal (3):
  - Novartis Investigative Site, Carnaxide - Linda-A-Velha, Lisbon District
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Cluj-Napoca, Jud Cluj, Romania
- Russia (7):
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Volzhskiy
- Spain (6):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Zaragoza
- Thailand (2):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Büyükçekmece / Ýstanbul
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Istanbul

REFERENCES:
- See also: The American Journal of Transplantation, Poster Abstracts, 2016 Provider: John Wiley & Sons, Ltd — https://doi.org/10.1111/ajt.13898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Full analysis set (24 month analysis)
Groups:
- Everolimus: Conversion from Calcineurin inhibitor (CNI) to everolimus in combination with Myfortic (mycophenolic acid) and steroids
- Standard CNI (Tac): Calcineurin inhibitor (CNI) continuation with Tacrolimus (Tac) in combination with Myfortic (mycophenolic acid), and steroids
- Standard CNI (CsA): Calcineurin inhibitor (CNI) continuation with Cyclosporine (CsA) in combination with Myfortic (mycophenolic acid) and steroids
Period: Completed Study Medication at Month 24
Arm/Group | Everolimus | Standard CNI (Tac) | Standard CNI (CsA)
Started | 353 (Randomized set - 360 Full analysis set - 353 Safety analysis set -346*) | 231 (Randomized set -231 Full analysis set -231 Safety analysis set -238**) | 125 (Randomized set-125 Full analysis set -125 Safety analysis set -121***)
Completed | 229 (completed at month 24) | 190 (completed at month 24) | 93 (completed at month 24)
Not Completed | 124 | 41 | 32
Not completed — Adverse Event | 87 | 18 | 17
Not completed — Abnormal laboratory value(s) | 6 | 0 | 1
Not completed — Abnormal test procedure result(s) | 3 | 0 | 1
Not completed — Lack of Efficacy | 2 | 1 | 2
Not completed — Subject's no longer required drug | 1 | 1 | 1
Not completed — Withdrawal by Subject | 18 | 8 | 2
Not completed — Lost to Follow-up | 1 | 4 | 2
Not completed — Administrative problems | 2 | 1 | 2
Not completed — Death | 2 | 1 | 2
Not completed — Graft loss | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 5 | 2
Not completed — Missing | 2 | 0 | 0
Period: Completed Study Phase at Month 24
Arm/Group | Everolimus | Standard CNI (Tac) | Standard CNI (CsA)
Started | 353 (It includes those discontinued treatment) | 231 (It includes those discontinued treatment) | 125 (It includes those discontinued treatment)
Completed | 313 (at month 24) | 215 (at month 24) | 111 (at month 24)
Not Completed | 40 | 16 | 14
Not completed — Withdrawal by Subject | 18 | 6 | 3
Not completed — Lost to Follow-up | 10 | 5 | 7
Not completed — Death | 8 | 5 | 4
Not completed — Other | 2 | 0 | 0
Not completed — Missing | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS), 24 month analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Standard CNI (Tac) | Standard CNI (CsA) | Total
Number analyzed (Participants) | 353 | 231 | 125 | 709
Age, Continuous [Mean (Standard Deviation); unit: years] — Kidney transplant Recipients age in years
  years | 46.0 (14.4) | 47.3 (14.5) | 45.4 (15.6) | 46.2 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 71 | 33 | 215
  Male | 242 | 160 | 92 | 494
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 246 (69.7) | 173 (74.9) | 97 (77.6) | 516
  Black | 4 (1.1) | 5 (2.2) | 0 (0) | 9
  Asian | 66 (18.7) | 41 (17.7) | 20 (16.0) | 127
  Native American | 1 (0.3) | 0 (0.0) | 0 (0.0) | 1
  Pacific Islander | 0 (0) | 1 (0.4) | 1 (0.8) | 2
  Other | 36 (10.2) | 11 (4.8) | 7 (5.6) | 54

OUTCOME MEASURES:

1. Primary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: Assessment of renal function by comparing change from randomization to Month 12 in eGFR (MDRD4) between treatment arms (Full analysis set). Renal function was assessed by estimated Glomerular Filtration Rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) formula. MDRD formula: GFR [mL/min/1.73m˄2] = 186.3*(C˄-1.154)*(A˄-0.203)*G*R. DEFINITIONS: C = serum concentration of creatinine [mg/dL]; A = age [years]; G = 0.742 when gender is female, otherwise G = 1; R = 1.21 when race is black, otherwise R = 1
Time Frame: Month 12
Population: Full Analysis set - observed eGFR values at month 12 (counted the patients with available values)
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Groups:
- Standard CNI (Tac): Calcineurin inhibitor (CNI) continuation with Tacrolimus (Tac) in combination with Myfortic (mycophenolic acid) and steroids
- Standard CNI (CsA): Calcineurin inhibitor (CNI) continuation with Cyclosporine (CsA) in combination with Myfortic (mycophenolic acid), and steroids
Arm/Group | Everolimus | Standard CNI (Tac) | Standard CNI (CsA)
Number analyzed (Participants) | 327 | 213 | 116
mL/min/1.73m^2 | 64.1 (22.31) | 61.5 (19.86) | 58.4 (19.62)

2. Secondary Outcome: Incidence of Composite Efficacy Endpoint for Each Arm at Month 12 and Month 24
Description: Efficacy failure rate used the composite endpoint of: (1) treated biopsy-proven acute rejection (BPAR)*, (2) graft loss**, or (3) death . *A treated BPAR was defined as a biopsy graded IA, IB, IIA, IIB, or III and which was treated with anti-rejection therapy. **Graft loss is defined as when the allograft was presumed lost on the day the participant started dialysis and was not able to subsequently be removed from dialysis or re-transplanted.
Time Frame: at 12 months and month 24 post-transplantation
Population: Full Analysis Set
Measure: Number; unit: Number of incidence
Arm/Group | Everolimus | Standard CNI (Tac) | Standard CNI (CsA)
Number analyzed (Participants) | 359 | 231 | 125
Number of incidence
  Month 12 | 21 | 4 | 8
  Month 24 | 27 | 8 | 8

3. Secondary Outcome: Change in Left Ventricular Mass Index (LVMi) From Randomization to Month 12 and Month 24
Description: Evolution of left ventricular mass and hypertrophy were evaluated by left ventricular mass index (LVMi) assessed by echocardiography. LVMi is derived using a standard formula from dimensional measurements on the echocardiogram. Analysis of covariance was applied with treatment, center (as a random effect), and donor type as factors and LVMi at Randomization as covariate.
Time Frame: Randomization, Month 12 and Month 24
Population: Full Analysis Set consists of only patients with triple LVMi values available at randomization, Month 12 and month 24 are included
Measure: Mean (Standard Deviation); unit: g/m^2.7
Arm/Group | Everolimus | Standard CNI (Tac) | Standard CNI (CsA)
Number analyzed (Participants) | 180 | 156 | 75
g/m^2.7
  Randomization | 50.30 (11.62) | 51.08 (14.11) | 51.13 (12.70)
  Month 12 | 49.95 (12.63) | 48.98 (14.63) | 50.96 (13.00)
  Month 24 | 46.66 (12.19) | 45.63 (13.50) | 47.91 (12.71)

4. Secondary Outcome: Comparison of Incidence Rates of Efficacy Endpoints Between Treatment Arms (Full Analysis Set - 24 Month Analysis)
Description: (treated BPAR ≥ IB, graft loss or death)A comparison of the incidence rates for the individual components of the composite efficacy endpoint between treatment arms
Time Frame: at 24 months post-transplantation
Population: Full Analysis Set
Measure: Number; unit: Number of incidence
Arm/Group | Everolimus | Standard CNI (Tac) | Standard CNI (CsA)
Number analyzed (Participants) | 353 | 231 | 125
Number of incidence
  Composite failure: tBPAR>=IB, graft loss, death | 27 | 8 | 8
  Composite tBPAR>=IB, graft loss, death, loss f/u | 35 | 14 | 15
  Composite of graft loss or Death | 10 | 6 | 4
  tBPAR>=IB | 18 | 3 | 5
  Graft loss | 4 | 2 | 2
  Death | 8 | 5 | 4
  Suspected Acute rejection | 61 | 27 | 19
  Subclinical Acute rejection | 0 | 0 | 0
  Acute rejection (AR) | 52 | 14 | 15
  Treated Acute rejection (tAR) | 40 | 9 | 14
  biopsy proven acute rejection (BPAR) | 37 | 8 | 13
  treated biopsy proven acute rejection (tBPAR) | 32 | 7 | 13
  tBPAR=IA | 16 | 3 | 8
  tBPAR=IB | 14 | 3 | 5
  tBPAR=IIA | 3 | 0 | 1
  tBPAR=IIB | 2 | 0 | 0
  tBPAR=III | 0 | 0 | 0
  Antibody tBPAR | 2 | 1 | 1
  Antibody mediated rejection (AMR) | 16 | 4 | 3

ADVERSE EVENTS:
Time Frame: 24 months
Description: Incidence of serious adverse events/infections by primary system organ class and preferred tem and treatment- Safety analysis set
Arm/Group | Everolimus | Standard CNI (Tac) | Standard CNI (CsA)
Serious Adverse Events (participants affected / at risk) | 188/346 | 118/238 | 58/121
Other Adverse Events (participants affected / at risk) | 316/346 | 216/238 | 103/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=346) | Standard CNI (Tac) (N=238) | Standard CNI (CsA) (N=121)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 3 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphocytic infiltration (Blood and lymphatic system disorders) | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 2
Cardiac failure (Cardiac disorders) | 4 | 2 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 15 | 9 | 4
Food poisoning (Gastrointestinal disorders) | 1 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Ileal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Death (General disorders) | 1 | 1 | 1
Device leakage (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 3 | 0
Pyrexia (General disorders) | 25 | 5 | 4
Sudden death (General disorders) | 2 | 0 | 0
Surgical failure (General disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Kidney transplant rejection (Immune system disorders) | 19 | 5 | 8
Transplant rejection (Immune system disorders) | 23 | 5 | 9
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0
BK virus infection (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1
Catheter site abscess (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0 | 0
Corona virus infection (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 4 | 4 | 3
Cytomegalovirus viraemia (Infections and infestations) | 1 | 1 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 11 | 9 | 5
Gastroenteritis norovirus (Infections and infestations) | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 3 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0
Graft infection (Infections and infestations) | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 2 | 0 | 0
Herpes simplex (Infections and infestations) | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 3 | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 2 | 0 | 0
Peritoneal tuberculosis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 14 | 4 | 5
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 13 | 4 | 5
Pyelonephritis acute (Infections and infestations) | 4 | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1
Renal cyst infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 1 | 0 | 0
Scrub typhus (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 6 | 0 | 1
Septic necrosis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Shunt infection (Infections and infestations) | 1 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0
Urinary tract infection (Infections and infestations) | 25 | 19 | 8
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 9 | 5 | 4
Vestibular neuronitis (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Zygomycosis (Infections and infestations) | 1 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Colon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 5 | 5 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 4 | 1
Graft loss (Injury, poisoning and procedural complications) | 2 | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal graft loss (Injury, poisoning and procedural complications) | 1 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 | 2 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 2 | 2 | 1
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Biopsy (Investigations) | 2 | 0 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0
Blood creatinine abnormal (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 17 | 6 | 5
C-reactive protein increased (Investigations) | 1 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Haemoglobin urine present (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 5 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Multifocal motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 5 | 3 | 1
Hydronephrosis (Renal and urinary disorders) | 3 | 2 | 1
Kidney fibrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephritis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 8 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 2 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 7 | 3 | 7
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 6 | 6 | 2
Renal tubular atrophy (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 4 | 1 | 1
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Urinary fistula (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 4 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 6 | 2 | 0
Haematoma (Vascular disorders) | 1 | 1 | 1
Haemodynamic instability (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0
Lymphocele (Vascular disorders) | 2 | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Necrosis ischaemic (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 2 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=346) | Standard CNI (Tac) (N=238) | Standard CNI (CsA) (N=121)
Anaemia (Blood and lymphatic system disorders) | 41 | 21 | 5
Leukopenia (Blood and lymphatic system disorders) | 48 | 35 | 11
Diarrhoea (Gastrointestinal disorders) | 79 | 55 | 13
Mouth ulceration (Gastrointestinal disorders) | 24 | 2 | 1
Nausea (Gastrointestinal disorders) | 21 | 14 | 4
Vomiting (Gastrointestinal disorders) | 21 | 9 | 3
Oedema peripheral (General disorders) | 60 | 21 | 13
Pyrexia (General disorders) | 62 | 20 | 12
Nasopharyngitis (Infections and infestations) | 31 | 23 | 10
Upper respiratory tract infection (Infections and infestations) | 20 | 19 | 2
Urinary tract infection (Infections and infestations) | 75 | 47 | 18
Blood creatinine increased (Investigations) | 30 | 24 | 20
Diabetes mellitus (Metabolism and nutrition disorders) | 15 | 19 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 26 | 11 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 40 | 15 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 17 | 11 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 13 | 1
Proteinuria (Renal and urinary disorders) | 52 | 11 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 16 | 3
Acne (Skin and subcutaneous tissue disorders) | 19 | 8 | 3
Hypertension (Vascular disorders) | 35 | 24 | 12
BK virus infection (Infections and infestations) | 5 | 13 | 5
Cytomegalovirus infection (Infections and infestations) | 13 | 13 | 9
Gastroenteritis (Infections and infestations) | 20 | 18 | 8
Pneumonia (Infections and infestations) | 20 | 8 | 6
Kidney transplant rejection (Immune system disorders) | 22 | 6 | 9
Transplant rejection (Immune system disorders) | 26 | 7 | 10
Hematuria (Renal and urinary disorders) | 15 | 18 | 2
Renal impairment (Renal and urinary disorders) | 17 | 13 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing any publications from a single-site are postponed until publication of the pooled data (i.e., data from all sites) in the clinical trial.